CLINICAL TRIAL: NCT04836897
Title: Evaluation of the Efficacy and Safety of the Transcatheter Aortic Valve Replacement System in Patients With Severe Aortic Valve Stenosis Disease at High Surgical Risk
Brief Title: PrizValve® Transcatheter Aortic Valve Replacement Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-valve-2020-07
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Transcatheter aortic valve replacement
  Interventions: Device: PrizValve® valve and transapical delivery system

INTERVENTIONS:
Device: PrizValve® valve and transapical delivery system — Transcatheter aortic valve replacement system

SUMMARY:
The purpose of this clinical study is to evaluate the effectiveness and safety of the transcatheter aortic valve system in the treatment of patients with severe aortic stenosis who are at high risk of surgery or who are not suitable for surgery.

DETAILED DESCRIPTION:
This study is an multicenter, single-arm, prospective, safety and performance clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years ;
2. Patients with symptomatic severe aortic valve stenosis (evaluated by echocardiography: transaortic valve pressure gradient ≥40mmHg (1mmHg=0.133kPa), or transaortic valve blood flow rate ≥4m/s, or aortic Valve area<1.0cm2, or AVA <0.5cm2 /m2);
3. NYHA ≥ II;
4. Life expectancy> 12 months;
5. Patients who are anatomically suitable for transcatheter aortic valve implantation;
6. After evaluation by two or more cardiovascular surgeons, patients who are unsuitable for surgery; or patients who refuse surgery after sufficient communication by the surgeons and are at high risk of routine surgery;
7. Patients who can understand the purpose of the trial, voluntarily participate in and signed informed consent form, and are willing to accept relevant examinations and clinical follow-ups.

Exclusion Criteria:

1. Acute myocardial infarction occurred within 1 month before this treatment;
2. Congenital single leaf aortic valve;
3. Any therapeutic cardiac operation (including placement of coronary drug-eluting stents) within 30 days;
4. The patient's heart has been implanted with other artificial heart valves, artificial rings, or severe mitral regurgitation (>3+);
5. Blood system diseases or abnormalities, including leukopenia (WBC<3×109/L), acute anemia (HB <90g/L), thrombocytopenia (PLT<50×109/L), bleeding constitution and coagulopathy ；
6. Untreated severe coronary artery stenosis that requires revascularization;
7. Patients with hemodynamic or respiratory instability, requiring continuous mechanical heart assistance or mechanical ventilation;
8. Patients who need emergency surgery for any reason;
9. Hypertrophic cardiomyopathy with obstruction;
10. Severe left ventricular dysfunction, left ventricular ejection fraction (LVEF) <20%;
11. The echocardiogram indicates the presence of a heart mass, thrombus or vegetation;
12. A history of acute peptic ulcer or upper gastrointestinal bleeding within 3 months;
13. Are allergic to cobalt-chromium alloys or contrast agents, and cannot tolerate anticoagulation and antiplatelet therapy;
14. The diameter of the aortic valve annulus <16mm or >28mm;
15. In any case, patients who refuse surgical treatment in emergency situations;
16. Cerebrovascular accident occurred within 3 months, not including transient ischemic attack;
17. Severe aortic diseases, including abdominal aortic or thoracic aortic aneurysm, obvious curvature of the aortic arch, atherosclerosis of the aortic arch, narrowing of the abdominal or thoracic aorta, and obvious curvature or extension of the thoracic aorta;
18. The iliac-femoral artery is severely obstructed with calcification, severely tortuous or unable to place the 1418F catheter sheath kit;
19. Active infective endocarditis or other active infections;
20. Aortic valve leaflets calcified plaque close to the coronary ostium;
21. Severe disability Alzheimer's disease and unable to take care of oneself in life;
22. Those who have participated in clinical trials of other drugs or medical devices before entering the group and have not yet reached the time limit of the primary research endpoint;
23. The researcher judged that the patient had poor compliance and could not complete the study as required.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Freedom from all-cause mortality | 12 months
  All-cause mortality within 12 months of TAVI procedure

SECONDARY OUTCOMES:
Freedom from all-cause mortality | 2-5 years
  All-cause mortality within 2-5 years of TAVI procedure
Device success | immediate post-surgical
  Device success after TAVI
Procedural success | immediate post-surgical
  Procedural success after TAVI
Rate of Myocardial infarction | 30 days、6 months、1-5 years
  Rate of Myocardial infarction after TAVI
Rate of All disabling stroke | 30 days、6 months、1-5 years
  Rate of All disabling stroke after TAVI
Rate of Severe bleeding | 30 days、6 months、1-5 years
  Rate of Severe bleeding after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Chen mao, Chief, Study Chair — Study Principal Investigator
Locations (1):
- Department of Cardiology, West China Hospital, Sichuan University, Sichuan, China

IPD SHARING:
Plan to Share IPD: No